CLINICAL TRIAL: NCT07088406
Title: A Multi-level Mother-daughter Physical Activity Intervention for Pre- Adolescent Latinas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01CA292783 (NIH); 1R01CA292783-01 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Family Communication; Parenting Behavior
Keywords: Physical Activity; Conmigo; Mother-daughter; Latina; Multilevel Intervention; healthy eating; fruit and vegetable intake; parenting; YMCA facilitators
MeSH Terms: conditions — Motor Activity | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collection team is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Experimental): 10-week PA promotion program
  Interventions: Behavioral: Physical Activity Promotion
- Healthy Eating Intervention (attention control program) (Active Comparator): 10-week health eating intervention
  Interventions: Behavioral: Healthy Eating

INTERVENTIONS:
Behavioral: Physical Activity Promotion — The Conmigo Physical Activity intervention involves the delivery of ten weekly sessions led by YMCA Facilitators supported by Drs. Arredondo and Ayala, Project Manager and student research assistants. Mothers and daughters (8-11 years old) will be invited to participate in ten in-person 2-hour sessions on topics such as PA parenting, communication, goal setting, etc. Mothers and daughters participate together in most activities, with small group breakouts where just mothers or just daughters have separate activities during some sessions. Each session includes didactic teaching, skill building (e.g. role plays), interactive discussions, 30 minutes of group PA, and goal-setting/review of previous goals. Overall, the activities are designed to promote increased physical activity and mediators to PA (family communication, parenting strategies, etc.). Each cohort will include 12-15 mother-daughter dyads.
  Other Names: Conmigo
  Arms: Physical Activity Intervention
Behavioral: Healthy Eating — The Healthy Eating intervention involves the delivery of 10 sessions by YMCA facilitators supported by Drs. Arredondo and Ayala, the Project Manager, and student research assistants. Mothers and daughters (8-11 years old) will be invited to participate in 10 2-hour in-person sessions that include both large and small group activities. Overall, the activities are designed to promote engagement in dietary behavioral strategies and parenting strategies across contexts and settings to promote fruit, vegetable and fiber consumption. Large and small groups activities include goal setting, implementation planning, homework activities, and focused discussion on mediators (e.g., family communication, parenting strategies) and moderators (e.g. acculturation). Each cohort will include 12-15 mother-daughter dyads.
  Arms: Healthy Eating Intervention (attention control program)

SUMMARY:
The goal of this Cluster Randomized Control Trial (RCT) is to learn if the mother-daughter intervention titled "Conmigo" can increase Latina preadolescents' physical activity (PA). The main objectives of the study are:

* To test the effectiveness of Conmigo on daughters' Moderate-to-Vigorous level PA (MVPA) over time
* To evaluate individual (e.g. mothers' MVPA) and family level (e.g. mother-daughter communication) mechanisms of change and their bidirectional effects

Researchers will compare the 10-week physical activity promotion intervention to a 10-week parallel intervention with emphasis on another health behavior (dietary intake) to see if there are differences in MVPA levels. We will enroll 216 Latina mother-daughter pairs at 18 elementary schools; each school will randomly receive the PA intervention or the control group program.

Mothers and daughters will attend 10 weekly sessions (2 hours each) at their elementary school, led by YMCA staff. Informed by social cognitive theory and family systems theory, the PA intervention sessions target family-level correlates of physical activity such as PA promotion parenting strategies (monitoring, role-modeling, etc.) and mother-daughter communication. Participants in the intervention group engage in weekly PA during sessions, discuss different topics each week, and set goals and receive PA homework during the week.

The investigators hypothesize that daughters participating in Conmigo will have higher minutes of device-assessed MVPA at M2 (post program), M3 (6 months post program), and M4 (12-months post program) compared to girls in the control condition.

DETAILED DESCRIPTION:
Fewer Latina girls in the United States (US) meet current physical activity (PA) guidelines, especially those from lower-income and less-acculturated backgrounds-contributing to long-standing health disparities. The pre-pubertal phase (ages 8-11) represents a critical window for PA interventions to prevent the sharp decline in activity levels that typically occurs during adolescence.

To address this need, we will conduct a two-arm cluster RCT in 18 schools serving Latina girls to evaluate Conmigo, a multilevel, mother-daughter PA intervention. This trial builds on prior formative work and a successful R21 pilot feasibility study, which demonstrated promising increases in moderate-to-vigorous physical activity (MVPA) among Latina mother-daughter dyads following a 10-week intervention.

The current study will recruit and randomize 216 mother-daughter dyads (girls aged 8-11) to either the 10-week Conmigo intervention or an attention-control program of similar duration and structure focused on dietary intake. Both programs will be delivered by trained YMCA staff in partnership with participating schools. Using a Hybrid Type 1 effectiveness-implementation design, we will assess both the effectiveness of the intervention and key implementation outcomes to inform future scale-up.

At the individual level, girls will participate in PA sessions and learn behavioral strategies to support daily PA habits. At the family level, mothers will also attend the intervention sessions and receive additional instruction focused on PA parenting practices and strengthening mother-daughter communication. Mothers are critical to shaping their daughters' PA through modeling, creating active opportunities, limiting sedentary behaviors, and providing encouragement and support. Importantly, parent-child influences are bidirectional meaning that daughters also shape parenting practices and mothers' own PA behaviors through their needs and feedback.

Girls' PA will be objectively measured using accelerometer devices worn by mothers and daughters at baseline, 3, 9, and 15 months. Secondary outcomes include PA parenting practices and mother-daughter communication, as well as mothers' PA. Focus groups and interviews with participants, school personnel, YMCA staff, and community partners will identify facilitators and barriers to implementation, mechanisms of change, and strategies for wider dissemination.

Specific Aims are to:

1. Test the effectiveness of Conmigo in increasing girls' MVPA over time;
2. Examine individual (e.g., mothers' MVPA) and family-level (e.g., communication, parenting practices) mechanisms and their bidirectional influences on behavior change;
3. Use qualitative and quantitative methods to evaluate implementation outcomes, including feasibility, fidelity, and scalability across community settings.

By partnering with 9 YMCAs and 18 schools, Conmigo aims to strengthen community capacity to deliver culturally tailored, evidence-based PA interventions. This work addresses critical gaps in the literature by focusing on Latina mother-daughter dyads, incorporating objective outcome measures and long-term follow-up, and advancing implementation science within community health promotion efforts.

ELIGIBILITY:
Inclusion Criteria (DAUGHTER):

* Self-identifying as Latina
* aged 8-11
* not currently meeting CDC's 2018 PA guidelines (60 min MVPA/day)
* attends an elementary school enrolled in the study
* speaks English or Spanish

Inclusion Criteria (MOTHER):

* Self-identifying as Latina
* primary female caregiver (living with her ≥4 days/week) of the daughter
* speaks English or Spanish
* both Mother & Daughter can attend weekly program activities for 10 weeks, and intend to stay in the area for the study's duration.

Exclusion criteria:

* either Mother or Daughter has a health condition that precludes them from doing PA
* cognitive impairment affecting participation,
* inability for mother to provide informed consent or daughter to provide assent in English or Spanish

Ages: 8 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mothers and daughters self-identifying as women
Enrollment: 432 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in daughters' objective PA | From enrollment to 3 months, 9 months, and 15 months
  Change in daughters' accelerometer-assessed minutes per day of moderate-to-vigorous physical activity (MVPA); worn for at least four 10+ hour days.

SECONDARY OUTCOMES:
Change in Mother-daughter communication | From enrollment to 3 months, 9 months, and 15 months
  Completed by Mothers; assessed by Parent Adolescent Communication Scale (PACS) -Open Family Communication Domain. 10 items on a 5-point likert scale of strongly disagree to strongly agree. Sum total score ranges from 10-50, with 50 representing more open (better) mother-daughter communication.
Change in Physical Activity Parenting Strategies | From enrollment to 3 months, 9 months, and 15 months
  Completed by mothers; assessed with two domains (Nondirective support and Guided Choice) of the Physical Activity Parenting Practices (PAPP) scale which assesses mothers' use of parenting strategies that promote physical activity (PA) among 5-12 year old children. Nondirective support is a 10-item scale; guided choice is a short-version 4-item scale. Participants respond on a 5-point likert scale of frequency which is scored 0-4 per item and sum totaled. Nondirective support subscores range from 0-40; Guided choice subscores range from 0-16. The total combined score from both domains ranges from 0-56 with a higher score meaning more frequent use of PA-promoting parenting strategies.
Change in Daughters' Dietary Intake | From enrollment to 3 months
  Completed by daughters (with mother's assistance); Block Yesterday food screener. This screener assesses children's intake by food group; the focus is on intake of fruit and fruit juices, vegetables, potatoes, whole grains, meat/poultry/fish, dairy, legumes, saturated fat, "added sugars", glycemic load and glycemic index. A secondary analysis produces estimates for intake of sugary beverages (both kcal and frequency). Screeners are externally analyzed by Nutrition Quest (https://www.nutritionquest.com/) with outcomes measured in number of servings consumed.
Change in Mother's Physical Activity | From enrollment to 3 months, 9 months, and 15 months
  Change in mothers' minutes per day of accelerometer-assessed moderate-to-vigorous physical activity; worn for at least four 10+ hour days.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Our data and resources generated by the study will include: (1) deidentified demographic and survey data; (2) physical activity tracking using accelerometers; (3) anthropometrics including height and weight; (4) study protocols (including analysis plans and consent forms); (6) training protocols; and (7) intervention materials.
  Codebooks and data collection instruments will also be made available to facilitate the interpretation of study findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available within 6 months of the study end and primary outcome paper publication. The data will be available for a minimum of 7 year following completion of the study in the repository.
Access Criteria: The scientific data and metadata from this project will be archived in the SDSU Institutional Repository and others, ensuring long-term preservation and accessibility.
  We will also share study protocols and training materials for community-based physical activity interventions and assessments. Some materials will be openly accessible through SDSU-affiliated portals, while deidentified datasets will be released upon request under a data-sharing agreement that provides for commitment to: (1) using the data only for research purposes, (2) to securing the data, and (3) to destroying or returning the data after analyses are completed. Data and intellectual property generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy.